CLINICAL TRIAL: NCT06522477
Title: Feasibility of High and Low Intensity Virtual Reality Gait Training in Individuals with Chronic Stroke: a Pilot Study
Brief Title: High Vs Low Intensity Virtual Reality Gait Training in Individuals with Chronic Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Christopher Henderson, Assistant Research Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23656
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Gait Disorders, Neurologic
Keywords: stroke; gait; rehabilitation; high-intensity; virtual reality
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to receive up to 15 visits/5 weeks of high- or low-intensity virtual reality gait training. Following a 4 week washout, they will complete the alternative intervention.
Who Masked: Outcomes Assessor
Masking Description: Blinded clinical assessors will perform assessments of clinical outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity followed by low-intensity virtual reality gait training (Experimental): Individuals randomized to this group will first perform high-intensity virtual reality gait training and following a 4-week washout period will complete low-intensity virtual reality gait training.
  Interventions: Other: Virtual reality gait training
- Low-intensity followed by high-intensity virtual reality gait training (Experimental): Individuals randomized to this group will first perform low-intensity virtual reality gait training and following a 4-week washout period will complete high-intensity virtual reality gait training.
  Interventions: Other: Virtual reality gait training

INTERVENTIONS:
Other: Virtual reality gait training — Individuals will walk on a treadmill with overhead harness system in place while viewing 1st-person perspective walking videos on a television placed immediately in front of the treadmill.

SUMMARY:
The purpose of this pilot study is to investigate the feasibility of 1) providing virtual reality walking training using a custom developed setup able to be replicated in routine clinical practice and 2) combining the virtual reality training with high-intensity gait training.

DETAILED DESCRIPTION:
This study will utilize a randomized-crossover design. Following confirmation of eligibility and completion of Baseline 1 testing, individuals will be randomized to receive up to 15 visits over approximately 5 weeks of either high or low intensity virtual reality gait training. Following which, individuals will undergo Post 1 testing to capture potential change in outcomes following the intervention. Participants will then take at least a 4-week break before returning to complete Baseline 2 testing and up 15 visits over 5 weeks of the alternative intervention before finally completing Post 2 testing.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral deficits following stroke > 6 months prior; however individuals > 4 months post-stroke are eligible for consenting, but final eligibility and potential enrollment will not occur until > 6 months
* Age 18-85 years
* Weight < 350 pounds
* Able to follow a 3-step command
* Able to ambulate with self-selected gait speeds between 0.01-1.0 m/s without physical assistance, but with below knee bracing and/or assistive device as needed
* Lower extremity Fugl-Meyer < 34
* Medical clearance to participate

Exclusion Criteria:

* Evidence of cerebellar ataxia
* Uncontrolled cardiopulmonary or metabolic disease that limits exercise participation, active heterotopic ossification, recurrent history of lower extremity fractures, previous orthopedic or other peripheral or central neurologic injury that may impair locomotor activities
* Currently participating in other physical therapy
* > 50 units of Botox in the lower extremity OR in the lower extremity, but above the knee if the participant wears an ankle-foot-orthosis (AFO) within the past three months. Note that participants may be consented prior to 3 months post-injection; however, eligibility will be determined post 3 months.
* Unable to read > 50% of the letters on the 20/70 line of the Snellen Chart with customary eye wear at a distance of 20 feet

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Gait speed | After 5 weeks of training
  This is an assessment of overground walking speed measured across a distance of ~20 feet and will be conducted at both self-selected (instructions: "walk at your usual, comfortable pace") and fastest (instructions: "walk as fast as you safely can") walking speeds.
6 minute walk test | After 5 weeks of training
  Individuals will be asked to "cover as much ground as possible" over a six minute period.
Peak treadmill speed | After 5 weeks of training
  Individuals will participate in a walking-based graded exercise test. While harnessed for safety on a treadmill, the treadmill will be initially set to 0.1 m/s and increased by 0.1 m/s each minute until the test is terminated due to one of the following: 1) the participant requests to stop, 2) the participant is unable to keep up with the speed of the treadmill and/or loses their balance, 3) any of the absolute exercise test termination criteria provided by American College of Sports Medicine are present. The highest speed that the individual can walk for a minute at is the peak treadmill speed.

SECONDARY OUTCOMES:
Mini Balance Evaluation Systems Test | After 5 weeks of training
  14 item assessment of static and dynamic balance. Example tasks include sit to stand, stand on one leg, standing stepping reactions, and walking with head turns.
Steps per Day | After 5 weeks of training
  Participants will wear a research-grade pedometer (StepWatch; Modus Health) during waking hours for ~1-2 weeks before beginning each training protocol and after completing training protocol to quantify home and community mobility.
30 second Sit to Stand Test | After 5 weeks of training
  Participants will be asked to rise from a chair without using their arms and then return to sitting as many times as possible in 30 seconds.
Activity-Specific Balance Confidence (ABC) Scale | After 5 weeks of training
  This questionnaire asks individuals to rate their balance-confidence from 0 (no confidence) to 100 (completely confident) during a variety of 16 commonly performed tasks such as walking around a house or getting into a car.
Medical Outcomes Survey Short-Form 36 (SF-36) | After 5 weeks of training
  This 36-question survey asks individuals about how their current health may limit their ability to perform typical physical and social activities. Scores range from 0 (negative health) to 100 (positive health).
Oxygen Consumption | After 5 weeks of training
  Oxygen consumption will be measured via a portable metabolic cart (K5; COSMED) during the previously described graded exercise test. Participant will wear a snug fitting mask that covers their mouth and nose, but does not affect the amount or quality of air that they breathe. The mask will be connected to a small backpack that collects information on the rate of breathing and oxygen consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Henderson, PhD, Principal Investigator — Indiana University
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after completion of study for 3 years